CLINICAL TRIAL: NCT03131583
Title: A Phase I, Single-Center, Open-Label, Single-Group Study to Evaluate Potential Pharmacodynamics of Drug-Drug Interaction Between SHR4640 and Febuxostat and Between SHR4640 and Colchicine in Patients With Gout
Brief Title: The Drug-Drug Interaction of SHR4640, Febuxostat and Colchicine in Patients With Gout
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR4640-103
Record Dates: First submitted 2017-02-27; First posted 2017-04-27 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Gout
Keywords: SHR4640 Febuxostat Colchicine pharmacodynamics
MeSH Terms: conditions — Gout | interventions — Colchicine; Febuxostat; ruzinurad

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort 1 (Experimental): Colchicine 0.5 mg Oral Tablet Day-14~Day16 qd, Febuxostat 80 mg Oral Tablet Day1 and Day8 qd, SHR4640 10 mg Oral Tablet Day3~Day8 qd.
  Interventions: Drug: Colchicine; Drug: Febuxostat; Drug: SHR4640

INTERVENTIONS:
Drug: Colchicine — Day-14~Day16 qd
Drug: Febuxostat — Day1 and Day8 qd
Drug: SHR4640 — Day3~Day8 qd

SUMMARY:
The objective of the study is to assess the pharmacodynamic properties of drug-drug of SHR4640, Febuxostat and Colchicine interaction in patients with gout.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a body mass index ≥18.5 and ≤30 kg/m2;
2. Screening sUA value ≥8mg/dl;
3. Subject has no clinically relevant abnormalities in vital signs, ECG, physical examination，imaging examination or safety laboratory values.

Exclusion Criteria:

1. Subject known or suspected of being sensitive to the study drugs or its ingredient；
2. sCr>ULN;
3. History of kidney stones or screening kidney stones by B-ultrasound；
4. History of malignancy within 5 years；
5. History of xanthinuria；
6. Donated blood（≥400ml）within 3 months prior to screening or received transfusion of blood。

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2018-01-29 (Actual); Study Completion 2018-01-29 (Actual)

PRIMARY OUTCOMES:
Maximun observed concentration (Cmax) of Febuxostat and Colchicine from plasma | Clinical significant changes from baseline up to Day 8
  PK profile
Area under the concentration-time curve (AUC) of Febuxostat and Colchicine from plasma | Clinical significant changes from baseline up to Day 8
  PK profile
Apparent terminal half-life (t1/2) of Febuxostat and Colchicine from plasma | Clinical significant changes from baseline up to Day 8
  PK profile

SECONDARY OUTCOMES:
Incidence of Adverse events | Clinical significant changes from Day-14 up to Day 16
  Safety issue
Changes in Laboratory Values | Clinical significant changes from Day-14 up to Day 16
  Safety issue
Changes in Electrocardiogram | Clinical significant changes from Day-14 up to Day 16
  Safety issue
Changes in Vital Signs Parameters | Clinical significant changes from Day-14 up to Day 16
  Safety issue

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No